CLINICAL TRIAL: NCT00614341
Title: A Phase IV Clinical Trial. Effect of Pulsing Electromagnetic Fields on Lower Extremity Diabetic Neuropathy: A Pilot, Open-Label Study
Brief Title: Effect of Pulsing Electrical Fields on Lower Extremity Diabetic Neuropathy: A Pilot, Open-Label Study
Acronym: DPN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedRelief (Industry)
Responsible Party: Margaret F. Fay, PhD, RN, CCRC, Director Medical-Regulatory Affairs, MedRelief, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 600-001
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Last update posted 2008-02-13 (Estimated); Status verified 2008-01

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: diabetes mellitus; neuropathy; distal symmetric polyneuropathy; pulsed electric fild
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1, 2 (Active Comparator): 1. Pulse MedRelief SE 55
  2. Continuous MedRelief SE 55
  Interventions: Device: MedRelief SE 55

INTERVENTIONS:
Device: MedRelief SE 55 — 4150 Hz signal continuous or pulse, high intensity, high modulation for 6 hours each night during treatment phase

SUMMARY:
To determine if pulsed electric field therapy reduces lower leg and foot pain associated with diabetic neuropathy and lessens the need for medication.

The MedRelief device sends a sub-threshold electric signal through the skin using electrodes as means of signal delivery. The signal or waveform, frequency and strength were created to match the characteristics of signals the body generates to help natural healing.

DETAILED DESCRIPTION:
A multi-center, randomized, open-label study involving 23 patients with chronic diabetic peripheral neuropathy meeting study entry criteria. Subjects will be randomly assigned to receive one of two treatments using an FDA cleared MedRelief device: (1) a MedRelief SE 55 device set on "pulsed" mode at 10 microsecond burst intervals 4150 Ha, or (2) a MedRelief SE 55 device set on "continuous" mode at 4150 Hz. Subjects will wear the device on target foot each night for a minimum of 6 hours over a two week (15 day treatment)period.

Subjects will complete a daily pain diary, medication form, and device use form. Subject global assessments and physician global assessments will occur at baseline, study visits Day 7, Day 15 and Day 21 (end of study).

Response to therapy will include pain reduction, improvement in sensation, improved response to vibratory stimulation and reduction of edema in study subjects.

ELIGIBILITY:
Inclusion Criteria:

* currently diagnosed with diabetes mellitus
* confirmed diagnosis of diabetic peripheral neuropathy
* age 18 years to 75 years
* both males and females are eligible for study participation
* HgA1c level under 9
* Physician confirmed stable glycemic control for 3 months prior to enrollment
* baseline pain level over previous month of 5
* willing to sign IRB approved consent and follow study visit requirements
* if female of childbearing age willing to undergo urine pregnancy test

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-05; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Pain reduction in diabetic patients with chronic diabetic neuropathy | Day 21

SECONDARY OUTCOMES:
Improvement in sensation and overall foot condition | Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Sprague, MD, Principal Investigator — Nephrology and Rheumatology Associates
Locations (1):
- Nephrology and Rheumatology Associates, Augusta, Georgia, United States